CLINICAL TRIAL: NCT01400100
Title: Changes in Pancreatic Texture After Single-shot Administration of 500 µg Octreotide in the Gastroduodenal Artery During Pancreatoduodenectomy - a Double-Blinded Randomized Controlled Trial
Brief Title: Effects of Intraarterial Octreotide on Pancreatic Texture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josef Hospital Bochum (Other)
Responsible Party: Principal Investigator, Orlin Belyaev, Dr. med. Orlin Belyaev, St. Josef Hospital Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4033-11
Record Dates: First submitted 2011-07-07; First posted 2011-07-22 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Pancreatic Fistula
Keywords: octreotide; intraarterial; pancreatic hardness; pancreatoduodenectomy; durometer; dynamometer
MeSH Terms: conditions — Pancreatic Fistula | interventions — Octreotide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octreotide (Experimental): Study patients receive after randomization a single shot of 5 mL 500 µg Octreotide in the gastroduodenal artery at the time of its transection.
  Interventions: Drug: Intraarterial application of Octreotide
- Control (Placebo Comparator): Control patients receive after randomization a single shot of 5 mL 0,9% NaCL solution in the gastroduodenal artery at the time of its transection.
  Interventions: Drug: sterile NaCl (sodium chloride) 0,9% solution

INTERVENTIONS:
Drug: Intraarterial application of Octreotide — 500 µg / 5 ml Octreotide is given as a single bolus injection in the gastroduodenal artery intraoperatively.
  Other Names: Sandostatin (Novartis Pharma, Switzerland); Bendatreotid; Octreo; Siroctid; Octreotid
  Arms: Octreotide
Drug: sterile NaCl (sodium chloride) 0,9% solution — a single intraarterial shot of 5 ml saline solution in the gastroduodenal artery
  Other Names: Sodium chloride 0,9% solution
  Arms: Control

SUMMARY:
The aim of the study is to test the hypothesis that intraarterial bolus application of 500 µg Octreotide in the gastroduodenal artery during the resectional phase of pancreatoduodenectomy in patients with soft pancreatic tissue hardens the texture of the pancreatic remnant.

A primary end-point of the study is a change in pancreatic texture.

A secondary end-point is the rate of postoperative pancreatic fistula.

DETAILED DESCRIPTION:
Soft pancreas is an established risk factor for the development of postoperative pancreatic fistula in patients undergoing pancreatoduodenectomy. Octreotide is believed to harden the pancreas. This theory is based on the results of a single animal experiment and a small case series in humans. This hardening effect of octreotide has not quantitatively been proven in humans and its mechanism is not clear. Histomorphologic correlates of pancreatic hardness are unknown.

In this study all patients who are eligible for pancreatoduodenectomy and sign the informed consent for participation in the study will be recruited. Those of them who prove to have a soft pancreas intraoperatively will receive a single bolus of 500 µg Octreotide in the gastroduodenal artery after its proximal division. Pancreatic hardness in the region of the resection margin will be quantitatively assessed by a Shore durometer before the intervention and at several time-points after it. The suture-holding capacity of pancreatic tissue at the resection margin will be quantitatively assessed by a dynamometer. Histomorphological features of pancreatic tissue will be characterized in details at the Institute of Pathology in order to define possible correlates of pancreatic hardness.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 an 90 years
* planned pancreatoduodenectomy
* signed informed consent
* pancreatic hardness equal or less than 40 SU as measured by durometer
* normal vascular anatomy of the hepato-pancreatic region

Exclusion Criteria:

* planned distal pancreatic resection
* planned non-resectional pancreatic surgery
* acute pancreatitis at the time of surgery
* pancreatic hardness before intervention higher than 40 SU as measured by durometer
* intraoperatively unstable patient
* intraoperative complications
* allergy towards octreotide
* anatomical variation of the vascular supply of the liver or pancreas posing an increased risk for octreotide distribution in other organs than pancreas
* lacking gastroduodenal artery or technically impossible cannulation of the artery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pancreatic hardness | 3 months postoperatively
  Pancreatic hardness is a quantifiable parameter, measured by a Shore Durometer in Shore Units on a 0-100 SU scale.

SECONDARY OUTCOMES:
Rate of postoperative pancreatic fistula | 3 months postoperatively
  Postoperative pancreatic fistula occurrs after pancreatoduodenectomy with an estimated rate of 5-30% depending on the definition used and a number of factors such as surgical technique, pancreatic texture, experience of the surgeon, hospital volume etc.

CONTACTS AND LOCATIONS:
Overall Officials: Orlin Belyaev, MD, Study Director — Department of Surgery, St. Josef Hospital; Christian Polle, Principal Investigator — Ruhr University of Bochum; Waldemar Uhl, MD, PhD, Study Chair — Department of Surgery, St. Josef Hospital
Locations (1):
- Department of Surgery, St. Josef Hospital, Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Foitzik T, Gock M, Schramm C, Prall F, Klar E. Octreotide hardens the pancreas. Langenbecks Arch Surg. 2006 Apr;391(2):108-12. doi: 10.1007/s00423-006-0030-z. Epub 2006 Mar 28. PMID 16568326
- [Background] Konstadoulakis MM, Filippakis GM, Lagoudianakis E, Antonakis PT, Dervenis C, Bramis J. Intra-arterial bolus octreotide administration during Whipple procedure in patients with fragile pancreas: a novel technique for safer pancreaticojejunostomy. J Surg Oncol. 2005 Mar 15;89(4):268-72. doi: 10.1002/jso.20193. PMID 15726611
- [Background] Belyaev O, Herden H, Meier JJ, Muller CA, Seelig MH, Herzog T, Tannapfel A, Schmidt WE, Uhl W. Assessment of pancreatic hardness-surgeon versus durometer. J Surg Res. 2010 Jan;158(1):53-60. doi: 10.1016/j.jss.2008.08.022. PMID 19394646
- [Derived] Belyaev O, Polle C, Herzog T, Munding J, Chromik AM, Meurer K, Tannapfel A, Bergmann U, Muller CA, Uhl W. Effects of intra-arterial octreotide on pancreatic texture: a randomized controlled trial. Scand J Surg. 2013;102(3):164-70. doi: 10.1177/1457496913490457. PMID 23963030